CLINICAL TRIAL: NCT01866969
Title: Physical, Emotional and Social Stressors and Their Impact on Quality of Life of Caregivers of Hospitalized Older Adults With Cancer
Brief Title: Quality of Life in Caregivers of Hospitalized Older Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13158; NCI-2013-01068 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13158 (Other: City of Hope Medical Center)
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2015-06

CONDITIONS: Hematopoietic/Lymphoid Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (quality of life questionnaire) (Experimental): Caregivers complete a self-administered questionnaire about factors associated with increased caregiver burden and decreased quality of life.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This clinical trial studies quality of life in caregivers of hospitalized older patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify patient and caregiver factors associated with increased caregiver burden and decreased quality of life in caregivers of older adults with cancer.

SECONDARY OBJECTIVES:

I. Determine characteristics of informal caregivers of older adults with cancer admitted to hospital.

II. Determine type and amount of care informal caregivers provide for older adults with cancer admitted to hospital.

III. Determine quality of life in informal caregivers of older adults with cancer admitted to hospital.

IV. Identify caregiver needs, both informational and resource related. V. Explore the association between re-admission to the hospital within 30 days and caregiver burden.

VI. Explore whether feedback of information attained from the assessment of the caregiver influences services implemented by the health care team.

VII. Determine reasons for non-participation.

OUTLINE:

Caregivers complete a questionnaire about their sociodemographics, physical health, social supports, social activity, mental health and caregiver burden. They will also provide an assessment of the person they care for.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Age >= 65 years old
* PATIENT: Diagnosis of cancer (solid or hematologic malignancy)
* PATIENT: Be able to provide informed consent
* PATIENT: Unplanned admission to hospital
* CAREGIVER: Primary caregiver (person who provides all of the majority of the unpaid care for the care recipient)
* CAREGIVER: Be able to provide informed consent

Exclusion Criteria:

* PATIENT: Planned admission to hospital for treatment (chemotherapy, transplant)
* CAREGIVER: Not fluent in English (because not all questionnaires have been validated in other languages)
* CAREGIVER: Paid and trained to care for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Caregiver burden and caregiver quality of life as measured by the Caregiver Quality of Life-Cancer Index | Up to 1 year
  Univariate analyses will be performed to test differences in the Caregiver Quality of Life-Cancer Index (CQOLC) total score and score of each domain (burden, distinctiveness, positive adaption, and financial concern) across categorical variables (analysis of variance [ANOVA]), and simple linear regression will be used to test association of CQOLC total score with continuous and categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Arti Hurria, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States